CLINICAL TRIAL: NCT01788215
Title: The Use of an MMP Inhibitor, Doxycycline, to Reduce Ovarian Androgen Production and Restore Normal Cycling in Women With Polycystic Ovarian Syndrome
Brief Title: Effect of a Commonly Used Antibiotic, Doxycycline, in Women With Polycystic Ovarian Syndrome
Acronym: MI-PCOS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Kathleen M. Hoeger, MD, Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RSRB 00034479
Record Dates: First submitted 2011-08-11; First posted 2013-02-11 (Estimated); Results first posted 2016-01-13 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2015-12

CONDITIONS: Polycystic Ovarian Syndrome (PCOS); Irregular Menstrual Cycles; Androgen Excess
Keywords: Polycystic Ovarian Syndrome; Irregular Menstrual Cycles; Androgen Excess in Women
MeSH Terms: conditions — Polycystic Ovary Syndrome; Menstruation Disturbances; Hyperandrogenism | interventions — Doxycycline; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Doxycycline (Active Comparator): Subjects randomized to receive doxycycline for a period of 12 weeks. A 12-week period thereafter will occur off study medication. The dose of doxycycline to be used in this study is 200mg/day in divided doses of 100mg twice daily. The dose of doxycycline being used in this study is 100mg because it is the standard approved dose.
  Interventions: Drug: doxycycline
- Sugar Pill (Placebo Comparator): The administered placebo is to be continued for a period of 12 weeks. A 12-week period thereafter will occur off placebo control
  Interventions: Other: Sugar Pill

INTERVENTIONS:
Drug: doxycycline — 200mg/day in divided doses of 100mg twice daily
  Arms: Doxycycline
Other: Sugar Pill — 1 pill twice a day
  Other Names: Placebo
  Arms: Sugar Pill

SUMMARY:
The purpose of this study is to study the effect of a commonly used antibiotic, doxycycline, on the production of ovarian hormones and menstrual cycles in women with Polycystic Ovarian Syndrome (PCOS).

DETAILED DESCRIPTION:
Polycystic ovarian syndrome (PCOS) is one of the leading causes of female infertility, affecting 5-10% of reproductive-age women . This heterogeneous disorder is characterized by anovulatory infertility, androgen excess, an increase in the ratio of LH to FSH, and morphologic polycystic changes to the ovaries. Obesity and insulin resistance are also metabolic factors associated with PCOS that further increase the morbidity in these patients. Inducing fertility in patients with PCOS can be a challenge, as it most often involves ovulation induction that can lead to ovarian enlargement, hyperstimulation, and multiple-birth pregnancies. This study is designed to determine novel effective strategies to promote normal cycling in this patient population.

ELIGIBILITY:
Inclusion Criteria:

1. Women between 18 and 40 years of age.
2. History of PCOS with < 8 periods the proceeding year
3. Clinical or biochemical evidence of androgen excess
4. BMI <40
5. Willingness to sign consent for study including participation with collection of blood specimens
6. Willingness to discontinue OCP for duration of study period up to 36 weeks

Exclusion Criteria:

1. Pregnancy
2. Hypersensitivity to doxycycline or tetracycline
3. History of Cushing's syndrome
4. History of hyperprolactinemia
5. History of congenital adrenal hyperplasia
6. Significant hepatic impairment, including serum AST or ALT >1.5 times upper limits of normal.
7. Significant renal impairment, GFR <60 ml/min
8. Current use of metformin, statins, glucocorticoids, spironolactone and/or anti-estrogens.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2010-11; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen M Hoeger, MD, MPH, Principal Investigator — University of Rochester; Stephen Hammes, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Strong Fertility Center, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 13 women were recruited. 3 did not meet inclusion/esclusion criteria.
Period: Overall Study
Arm/Group | Doxycycline | Sugar Pill
Started | 5 | 5
12 Weeks of Doxycycline or Placebo | 5 | 5
Completed | 3 | 4
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lost to Follow-up | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Doxycycline | Sugar Pill | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 10
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10
total serum testosterone [Mean (Standard Deviation); unit: ng/dL] | 50.6 (8.2) | 49.6 (8.2) | 50.1 (8.2)
free serum testosterone [Mean (Standard Deviation); unit: pg/mL] | 1.14 (0.57) | 1.36 (0.39) | 1.25 (0.48)
serum hormone binding globulin (SHBG) [Mean (Standard Deviation); unit: nmol/L] | 55.0 (13.2) | 44.0 (13.5) | 49.5 (13.4)

OUTCOME MEASURES:

1. Primary Outcome: Total Serum Testosterone
Description: We will determine total serum testosterone levels in all participating subjects at week 24.
Time Frame: 24 weeks
Population: in the sugar pill arm one participant dropped out at week 12
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Doxycycline | Sugar Pill
Number analyzed (Participants) | 5 | 4
ng/dL | 61.8 (13.6) | 41.6 (9.8)

2. Secondary Outcome: Serum Progesterone Levels in Blood
Description: Serum progesterone levels will be obtained on a weekly basis to assess ovulation. We will then perform statistical analysis on this data to determine the effectiveness of doxycycline in this study population.
Time Frame: 24 weeks
Population: This measurement was not completed, because the number of ovulations was measured in its place and better indicates the effect of the treatment. See outcome measure number 8.
Arm/Group | Doxycycline | Sugar Pill
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Total Serum Testosterone
Description: We will determine total serum testosterone levels in all participating subjects at week 12.
Time Frame: week 12
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Doxycycline | Sugar Pill
Number analyzed (Participants) | 5 | 5
ng/dL | 49.4 (10.8) | 43.0 (8.6)

4. Secondary Outcome: Free Testosterone in Serum
Time Frame: week 12
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Doxycycline | Sugar Pill
Number analyzed (Participants) | 5 | 5
pg/mL | 1.12 (0.39) | 1.16 (0.25)

5. Secondary Outcome: Free Testosterone in Serum
Time Frame: week 24
Population: in the sugar till arm, one participant dropped out at week 12
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Doxycycline | Sugar Pill
Number analyzed (Participants) | 5 | 4
pg/mL | 1.76 (1.56) | 1.08 (0.27)

6. Secondary Outcome: Serum Hormone Binding Globulin (SHBG)
Time Frame: week 12
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Doxycycline | Sugar Pill
Number analyzed (Participants) | 5 | 5
nmol/L | 50.4 (12.4) | 39.4 (10.9)

7. Secondary Outcome: Serum Hormone Binding Globulin (SHBG)
Time Frame: week 24
Population: in the sugar pill arm, one participant withdrew at week 12
Measure: Mean (Standard Deviation); unit: nmol /L
Arm/Group | Doxycycline | Sugar Pill
Number analyzed (Participants) | 5 | 4
nmol /L | 44.8 (10.6) | 36.2 (6.75)

8. Secondary Outcome: Total Number of Ovulations
Description: The total number of ovulations per group. Ovulation was defined as elevation of serum progesterone and or urinary pregnanediol glucuronide followed by documented menstrual bleeding within 2 weeks of elevation.
Time Frame: week 24
Population: In the sugar pill arm, one participant withdrew at week 12.
Measure: Number; unit: ovulations
Arm/Group | Doxycycline | Sugar Pill
Number analyzed (Participants) | 5 | 4
ovulations | 12 | 7

ADVERSE EVENTS:
Arm/Group | Doxycycline | Sugar Pill
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5

LIMITATIONS AND CAVEATS:
This study was underpowered due to reduced enrollment. Targeted enrollment was 40 and actual enrollment was 10.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes